CLINICAL TRIAL: NCT06904131
Title: A Phase I Clinical Trial of MUC1-targeted CAR-T Cells with PD1 Nanobody MSLN Dual-target for Advanced Gynecological Solid Tumors
Brief Title: A Phase I Clinical Trial of CAR-T Cells for Advanced Gynecological Solid Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Obstetrics & Gynecology Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUOBGY-2025-39
Record Dates: First submitted 2025-03-10; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Gynecological Solid Tumors
MeSH Terms: interventions — Cell- and Tissue-Based Therapy; Antibodies, Bispecific

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cell therapy group (Experimental): Screening patients who meet the criteria for peripheral blood mononuclear cell (PBMC) isolation and cell preparation. Based on the cell preparation status and mutual agreement between the researcher and the participant, the date of reinfusion (Day 0) is determined. On Days -5 to -3, the participant receives a conditioning regimen with cyclophosphamide and antithymocyte globulin. After recovery for two days (Days -2 and -1), on Day 0, the participant receives reinfusion of BZE2203 (dose determined according to the dose-escalation requirements). The safety observation period lasts for 28 days, and clinical efficacy is evaluated from Day 28 to Day 34. After comprehensive judgment, the second course of cell therapy is selected. Follow-up observations and evaluations are conducted once every three months, with follow-up visits once a year and telephone follow-ups once every two months.
  Interventions: Drug: Cell therapy with bispecific antibodies

INTERVENTIONS:
Drug: Cell therapy with bispecific antibodies — The dose-escalation phase is designed with three predefined dose levels, following a "3+3 design" and progressing from low to high doses. The "3+3" dose-escalation scheme is as follows: if no dose-limiting toxicity (DLT) occurs in the three subjects at a given dose level during the observation period, the dose will be escalated to the next higher level. If one subject out of the initial three experiences DLT at a dose level, an additional three subjects will be enrolled at that dose level for further DLT observation. The dose level at which no more than one subject out of the final six subjects experiences DLT will be defined as the maximum tolerated dose (MTD).

SUMMARY:
Screening patients who meet the criteria for peripheral blood mononuclear cell (PBMC) isolation and cell preparation. Based on the status of cell preparation and mutual agreement between the researcher and the participant, the date of reinfusion (Day 0) is determined. From Day -5 to Day -3, the participant receives a conditioning regimen with cyclophosphamide and antithymocyte globulin. After recovery for two days (Day -2 and Day -1), on Day 0, the participant receives reinfusion of BZE2203 (dose determined according to the dose-escalation requirements). The safety observation period lasts for 28 days, and clinical efficacy is assessed from Day 28 to Day 34. After comprehensive judgment, the second course of cell therapy is selected. Follow-up observations and evaluations are conducted once every three months, with follow-up visits once a year and telephone follow-ups once every two months.

DETAILED DESCRIPTION:
This study is a single-arm, open-label, dose-escalation and expansion clinical trial. The study is divided into two phases: the dose-escalation phase and the dose-expansion phase.

The dose-escalation phase is designed with three predefined dose levels, following a "3+3 design" and progressing from low to high doses. The "3+3" dose-escalation scheme is as follows: if no dose-limiting toxicity (DLT) occurs in the three subjects at a given dose level during the observation period, the dose will be escalated to the next higher level. If one subject out of the initial three experiences DLT at a dose level, an additional three subjects will be enrolled at that dose level for further DLT observation. The dose level at which no more than one subject out of the final six subjects experiences DLT will be defined as the maximum tolerated dose (MTD).

The dose level for the expansion phase will be determined based on a comprehensive consideration of the occurrence of DLT and the efficacy results obtained, with the actual occurrence serving as the basis.

The safety of CAR-T therapy will be assessed by monitoring adverse events (AE) following cell therapy. The efficacy of CAR-T therapy will be evaluated by observing disease response following cell therapy. Blood samples will be collected before cell infusion and within one year after infusion to measure the number of CAR-T cells, CAR copy number, and PD-1 nanobody concentration, thereby evaluating the pharmacokinetics of CAR-T cells. Blood samples will also be collected before cell infusion and within 28 days after infusion to measure the concentrations of relevant cytokines, in order to assess the pharmacodynamic characteristics of CAR-T therapy.

During the study, blood samples used for the production of CAR-T cells will be transported to Shanghai Cell Therapy Group Pharmaceutical Technology Co., Ltd. After the production of CAR-T cells is completed, the cells will be shipped to the study sponsor, who will then infuse the CAR-T cells into the corresponding subjects.

ELIGIBILITY:
inclusion criteria

1. Patients with gynecological solid tumors diagnosed by histopathology, with tumor tissue sample MUC1 expression rate ≥50% or MSLN expression rate ≥50%, PD-L1 positive expression, and sample source within 2 years;
2. Patients with advanced gynecological solid tumors who have failed standard treatment or are intolerant to such treatment and have no standard effective treatment options;
3. Females aged 18 to 70 years (inclusive);
4. Estimated survival time ≥ 3 months;
5. ECOG performance status score of 0 to 1 at screening and baseline;
6. Good organ and bone marrow function:

   1. The researcher assesses sufficient bone marrow function to receive lymphocyte-depleting chemotherapy: Neutrophil count ≥1.5 × 10^9/L, lymphocyte count ≥0.5 × 10^9/L;
   2. Platelet count ≥90 × 10^9/L;
   3. Hemoglobin ≥90 g/L (no blood transfusion or no erythropoietin-dependent within 7 days);
   4. Total bilirubin ≤2 times the upper limit of normal value;
   5. Serum creatinine ≤1.5 times the upper limit of normal value;
   6. Transaminase (AST, ALT) ≤2.5 times the upper limit of normal value (if liver metastasis is present, 5 times the upper limit of normal value);
   7. International Normalized Ratio (INR) or prothrombin time (PT) ≤1.5 times the upper limit of normal value;
   8. Pulmonary function: ≤ CTCAE grade 1 dyspnea and SaO2 ≥ 91% in room air;
   9. Cardiac function: Echocardiogram or radionuclide ventriculography (MUGA) assessment left ventricular ejection fraction (LVEF) ≥50% within 1 month of enrollment.

exclusion criteria

1. Participants who have undergone other anti-tumor treatments not allowed by the protocol within 1 month before CAR-T infusion (including radiotherapy, chemotherapy, small molecules, biological treatment, or immunotherapy, other research drugs);
2. Participants who have previously received targeted therapy against MUC1 or MSLN, or cellular therapy, or any gene therapy products (including CAR-T cell therapy) or any T cell therapy at home or abroad;
3. Pregnant or breastfeeding women;
4. AIDS virus, syphilis seroreactivity positive; hepatitis B surface antigen positive, or hepatitis B core antibody positive and hepatitis B virus DNA copies higher than the detection limit or greater than or equal to 1000 copies/mL; or hepatitis C virus infection;
5. Any uncontrollable active infection, coagulopathy, or any other major disease;
6. Patients with active autoimmune diseases being treated, organ transplantation and other immune-related diseases, or long-term use of immunosuppressive drugs such as glucocorticoids: a. Glucocorticoids cannot be discontinued within 72 hours before CAR-T cell infusion; b. Immunosuppressive agents other than glucocorticoids cannot be discontinued ≥4 weeks before enrollment;
7. Patients with severe cardiopulmonary insufficiency, uncontrolled hypertension, any of the following cardiovascular disease histories within the past 6 months: III or IV heart failure defined by the New York Heart Association (NYHA), cardiac catheterization or stent, myocardial infarction, unstable angina, or other clinically significant heart disease;
8. Patients with confirmed brain metastasis, or those with a history of or current central nervous system disease, such as epileptic seizures, cerebrovascular ischemia/hemorrhage, dementia, encephalopathy, or any autoimmune disease associated with the central nervous system;
9. Patients with high risk of bleeding or perforation;
10. Patients who underwent major surgery or significant trauma within 4 weeks before single collection;
11. Patients with other malignant tumors within 3 years or concurrently (except for skin basal cell carcinoma, cervical/breast cancer in situ, etc.);
12. Any other conditions deemed unsuitable for participation in the study by the investigator.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-11 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | The time frame was from subject enrollment until one year after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: XIN WU, chief physician, Study Director — Fudan University
Locations (1):
- The Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality, China